# LEAK AFTER SLEEVE GASTRECTOMY WITH POSITIVE INDOCYANINE GREEN TEST: AVOIDABLE SCENARIO?

RUNNING HEADS: Indocyanine green test for evaluation of perfusion of staple line of the stomach during laparoscopic sleeve gastrectomy

#### **AUTHORS:**

GIOVANNA PAVONE<sup>1</sup>, NICOLA TARTAGLIA<sup>1</sup>, MARIO PACILLI<sup>1</sup>, FRANCESCA MADDALENA<sup>1</sup>, FABIO PETRUZZELLI<sup>1</sup>,GENNARO MARTINES<sup>2</sup>, MICHELE DE FAZIO<sup>2</sup>, , ANTONIO AMBROSI<sup>1</sup>,.

# **AUTHORS:**

GIOVANNA PAVONE<sup>1</sup> MD, giovanna.pavone@unifg.it, DEPARTMENT OF MEDICAL AND SURGICAL SCIENCES, UNIVERSITY OF FOGGIA, VIALE PINTO, 71122, FOGGIA, ITALY. NICOLA TARTAGLIA<sup>1</sup> Prof. FACS,nicola.tartaglia@unifg.it, DEPARTMENT OF MEDICAL AND SURGICAL SCIENCES, UNIVERSITY OF FOGGIA, VIALE PINTO, 71122, FOGGIA, ITALY

MARIO PACILLI<sup>1</sup> MD, mario.pacilli@unifg.it, DEPARTMENT OF MEDICAL AND SURGICAL SCIENCES, UNIVERSITY OF FOGGIA, VIALE PINTO, 71122, FOGGIA, ITALY.

FRANCESCA MADDALENA¹ MD,<u>franc.maddalena@gmail.com</u>, DEPARTMENT OF MEDICAL AND SURGICAL SCIENCES, UNIVERSITY OF FOGGIA, VIALE PINTO, 71122, FOGGIA, ITALY.

FABIO PETRUZZELLI¹ MD, fabpetruzzelli33@gmail.com, DEPARTMENT OF MEDICAL AND SURGICAL SCIENCES, UNIVERSITY OF FOGGIA, VIALE PINTO, 71122, FOGGIA, ITALY. GENNARO MARTINES² Prof., gerrymartines@virgilio.it, DEPARTMENT OF GENERAL SURGERY AND LIVER TRANSPLANTATION, UNIVERSITY OF BARI, 70124 BARI, ITALY. MICHELE DE FAZIO² Prof., michele.defazio@uniba.it, DEPARTMENT OF GENERAL SURGERY AND LIVER TRANSPLANTATION, UNIVERSITY OF BARI, 70124 BARI, ITALY. ANTONIO AMBROSI¹ Prof., antonio.ambrosi@unifg.ti, DEPARTMENT OF MEDICAL AND SURGICAL SCIENCES, UNIVERSITY OF FOGGIA, VIALE PINTO, 71122, FOGGIA, ITALY.

## **AFFILIATIONS:**

1: DEPARTMENT OF MEDICAL AND SURGICAL SCIENCES, UNIVERSITY OF FOGGIA, VIALE PINTO, 71122, FOGGIA, ITALY.

2:DEPARTMENT OF GENERAL SURGERY AND LIVER TRANSPLANTATION "M. RUBINO", UNIVERSITY OF BARI, 70124 BARI, ITALY.

# CORRESPONDING AUTHOR:

NICOLA TARTAGLIA, <u>nicola.tartaglia@unifg.it</u>, Viale Pinto 1, 71122 Foggia, Italy tel./fax +39 0881.733808

Date Document: 30/03/2022

#### ABSTRACT

BACKGROUND: The staple line gastric leak (GL) is estimated to be the most serious complication of the sleeve gastrectomy. The use of indocyanine green (ICG) has been introduced in minimally invasive surgery to showthe vascularization of the stomach in real time and its application to the gastroesophageal junction (GE) during Laparoscopic Sleeve Gastrectomy (LSG) seems very promising.

CASE PRESENTATION: We present the case of a 40-year-old female underwent laparoscopic sleeve gastrectomy. Intraoperative indocyanine green test showed a small dark area in the proximal third of the staple line reinforced with fibrin glue. Two weeks later the patient presented to the emergency room (ED) with abdominal pain, fever, vomiting, intolerance to oral intake and the evidence of a leak on the abdomen Computer Tomography (CT).

CONCLUSIONS: This case report shows that intraoperative ICG test can be helpful in determining which patients are at greater risk of the leak and, more importantly, the cause of the leak but further tests are needed to determine if the ICG predicts leak due to ischemia.

Key words: laparoscopic sleeve gastrectomy, Indocyanine green test, gastric fistula.

# INTRODUCTION

Obesity is a major current public health problem of global significance. Obesity is associated with a myriad of serious health conditions, including hypertension, type II diabetes mellitus, sleep disorders, dementia, cardio-vascular diseases, and various malignancies, and is associated with increased morbidity and mortality [1].

Laparoscopic sleeve gastrectomy (LSG) has become in the last decades the most frequently performed bariatric procedure worldwide since it is a less demanding procedure compared to Roux-en-Y gastric bypass (BRGY), with a shorter operative time and absence of anastomosis. [2]

The staple line gastric leak (GL) is estimated to be the most serious complication of this procedure, due to a difficult healing process when using a non-standardized endoscopic approach, with a currently reported rate of 0.4 to 2.7%. [3]

Post LSG leaks can be misdiagnosed, resulting in delayed management and catastrophic consequences [4,5]. The clinical presentation, signs, and symptoms are highly variable, ranging from asymptomatic to septic shock [6].

Fistulas are complex and have multifactorial origins. Situations that cause difficulty in gastric emptying, with a consequent increase in intraluminal pressure, may lead to a rupture of the stapling line in the region of the esophagogastric junction, at the His angle, causing a gastric fistula [7]. Stapling failures, gastric twist, tissue damage, and distal strictures are some of the conditions that pose an additional risk for the development of fistulas after SG [8, 9].

The use of indocyanine green (ICG) has been introduced in minimally invasive surgery[10-12].

Indocyanine Green (ICG) is a liquid that can be injected into the human bloodstream without adverse effects. [13] The ICG fluoresces when excited with light of wavelength in the near infrared (NIR) spectrum (approximately 820 nm) [14] [15, 16]. Special telescopes detect the fluorescence that is transmitted to a standard monitor that allows the identification of the anatomical structures in which the dye is present (eg biliary tract, vessels, lymph nodes, etc.). It is a low cost technique capable of showing the

vascularization of the stomach in real time and its application to the gastroesophageal junction (GE) during LSG seems very promising [17-19].

In this article, we present a case report of a 40-year-old female with a positive intraoperative indocyanine green test as a prediction of the leak after sleeve gastrectomy.

#### CASE PRESENTATION

A 40-year-oldfemale with a body mass index of 43,1 Kg/m² and weighing 115 Kg underwent laparoscopic sleeve gastrectomy. Her past medical history includes hypertension, hypothyroidism with Basedow's disease, left eye glaucoma, depressive disorder. During the operation after four port placement, detachment from the great curvature with dissection of the gastroepiploic and short gastric vessels was performed employing an energy device.

The sleeve resection was shaped around a 40-French bougie in place using a mechanical linear stapler; 5 ml of ICG were then injected intravenously to identify the stomach, carefully assessing the angle of His (preoperative written informed consent was obtained from the patient).

Adequate perfusion was defined as "the direct and clear visualization of the fluorescence around the gastric tube, after an estimated time of 150-180 s following i.v. administration".

Intraoperative indocyanine green test showed a small dark area at the proximal third of the staple line, therefore it was decided to reinforce the suture line using fibrin glue (Figure 1a - 1b).

She had a smooth recovery with discharge home on the second postoperative day after a negative Gastrografin swallow test (Figure 2).

Two weeks later the patient presented to emergency department (ED) with abdominal pain, fever, vomiting and intolerance to oral intake. Her laboratory workups were within normal, computed tomography (CT) abdomen with oral and intravenous (IV) contrast revealed a collection 13x9 cm with air pocket adjacent to the staple line at the upper stomach (Figure 3).

The collection was treated with the placement of two abdominal drainages with laparoscopic approach and a self-expanding covered prosthesis placed with endoscopic technique to exclude the fistula (Figure 4-5). The patient was discharged in good general conditions, normal laboratory tests, control CT showing a clear reduction of the intra-abdominal collection (Figure 6). The patient will undergo a replacement of the prosthesis in 3/4 weeks.

#### DISCUSSION

The esophagogastric junction represents an anatomical area of weakness for any digestive suture. The fundic wall is thinner, and vascularization is more precarious than the rest of the stomach. This area under the cardia is more sensitive to technical failure or to any increase in intragastric pressure [20]. Experience showed us that almost all leaks after bariatric surgery originate in this location, namely just below the GE junction [21].

The gastric leakage could be due to the creation of a long and narrow tube with the maintenance of the pylorus which surely increases the intraluminal pressure (intragastric hypertension) or to the localized ischemia related to the gastroepiploic and the ligation of the short gastric vessel during the detachment a greater curvature or even an inadequate and abnormal inflammatory response to the surgical procedure [22, 23].

Recently, much interest has been focused on the possibility of assessing blood supply during surgery with the use of ICG fluorescence angiography, which is a real-time, inexpensive and feasible method of establishing vascularity in an selected area. [24,25]. It has been fully and positively approved in most laparoscopic procedures [26] but there is still little literature on its usefulness in bariatric procedures.

Di Furia et al. led a study on 43 patientsand concluded that intraoperative view of the blood supply of the stomach does not appear to represent a prognostic factor for the risk of gastric leakage, suggesting a complex multifactorial etiology (intragastric hypertension? Abnormal inflammatory response?) Which needs further data to be established[27].

Ortega et al. have obtained satisfactory results on 86 patients showing that ICG fluorescence angiography allows to determine the increased blood supply to the proximal stomach before any dissection during sleeve gastrectomy, so that an effort can be made to avoid unnecessary injury to these vessels during the procedure [28, 29]. Frattini et al. in their preliminary experience, the results of the ICG resemble the intraoperative methylene blue test and the postoperative contrast swallow test. The ICG allows for real-time assessment and provides a direct picture of tissue perfusion and vascularity. Furthermore, IGF may be useful in explaining the exact pathogenesis of gastric leak [30].

## **CONCLUSIONS**

Intraoperative ICG test can be helpful in determining which patients are at greater risk of the leak and, more importantly, the cause of the leak. In this case the fibrin glue was not sufficient to avoid the gastric fistula, but other reinforcement methods could be implemented in case of inadequate perfusion found with the ICG test, such as sutures. Further tests are needed to determine if the ICG predicts leak due to ischemia.

## REFERENCES

- 1. Van Gaal LF, Maggioni AP. Overweight, obesity, and out- comes: fat mass and beyond. Lancet (London, England). 2014;383:935–6.
- 2. .Hendricks L, Alvarenga E, Dhanabalsamy N, et al. Impact of sleeve gastrectomy on gastroesophageal reflux disease in a morbidly obese population. Undergoing bariatric surgery. Surg ObesRelat Dis. 2016;12:511–7.
- 3. Jung JJ, Jackson T, Gordon L, Hutter MM. Intraoperative leak test is associated with lower postoperative bleed rate in primary sleeve gastrectomy: a propensity matched analysis of primary and revision bariatric surgery using the MBSA- QIP database. SurgEndosc. 2021. https://doi.org/10.1007/s00464-020-08264-2.
- 4. Al Zoubi M, Khidir N, Bashah M. Challenges in the Diagnosis of Leak After Sleeve Gastrectomy: Clinical Presentation, Laboratory, and Radiological Findings. Obes Surg. 2021 Feb;31(2):612-616. doi: 10.1007/s11695-020-05008-y. Epub 2020 Oct 6. PMID: 33025538; PMCID: PMC7847981.

- 5. Sakran N, Goitein D, Raziel A, et al. Gastric leaks after sleeve gastrectomy: a multicenter experience with 2,834 patients. SurgEndosc. 2013;27(1):240–5. https://doi.org/10.1007/s00464-012- 2426-x.
- 6. Nedelcu M, Skalli M, Delhom E, et al. New CT scan classification of leak after sleeve gastrectomy. ObesSurg. 2013;23(8):1341–3. https://doi.org/10.1007/s11695-013-1002-3.
- 7. Yehoshua RT, Eidelman LA, Stein M, et al. Laparoscopic sleeve gastrectomyvolume and pressure assessment. Obes Surg. 2008;18(9):1083
- 8. Ferraz ÁAB, da Silva JD, Santa-Cruz F, et al. The impact of the gastric twist on esophagitis progression after sleeve gastrectomy: mid-term endoscopic findings. Obes Surg. 2020;30(11):4452
- 9. AbouRached A, Basile M, El Masri H. Gastric leaks post sleeve gastrectomy:review of its prevention and management. World J Gastroenterol. 2014;20(38):13904
- 10. Boni L, David G, Mangano A, et al. Clinical applications of indocyanine green (ICG) enhanced fluorescence in laparoscopic surgery. SurgEndosc. 2014. doi:10.1007/s00464-014-3895-x.
- 11. Pacilli M, Tartaglia N, Gerundo A, Pavone G, Fersini A, Ambrosi A. Energy Based Vessel Sealing Devices in Thyroid Surgery: A Systematic Review to Clarify the Relationship with Recurrent Laryngeal Nerve Injuries. Medicina (Kaunas). 2020 Nov 27;56(12):651. doi: 10.3390/medicina56120651. PMID: 33260912; PMCID: PMC7760641
- 12. Tartaglia N., Pavone G., Petruzzelli F., Di Lascia A., Vovola F., Maddalena F., Cianci P., Fersini A., Pacilli M., Ambrosi A. Robotic sleeve gastrectomy vs laparoscopic sleeve gastrectomy: ourpreliminaryexperience and a literaturereview. Clinical and Experimental Surgery. Petrovsky Journal. 2020; 8 (4): 7–15. DOI: https://doi.org/10.33029/2308-1198-2020-8-4-7-15
- 13. Alander JT, Kaartinen I, Laakso A, Pa ïtila T, Spillmann T, Tuchin VV, Venermo M, Valisuo P (2012) A review of indocyanine green fluorescent imaging in surgery. Int J BiomedImaging 2012:940585

- 14. Luo S, Zhang E, Su Y, Cheng T, Shi C (2011) A review of NIR dyes in cancer targeting and imaging. Biomaterials 32:7127–7138 15. Daskalaki D, Fernandes E, Wang X, Bianco FM, Elli EF, Ayloo S, Masrur M, Milone L, Giulianotti PC (2014) Indocyanine green (icg) fluorescent cholangiography during robotic cholecystectomy: results of 184 consecutive cases in a single institution. SurgInnov. doi:10.1177/1553350614524839
- 15. Spinoglio G, Priora F, Bianchi PP, Lucido FS, Licciardello A, Maglione V, Grosso F, Quarati R, Ravazzoni F, Lenti LM (2012) Real-time near-infrared (NIR) fluorescentcholangiography in single-site roboticcholecystectomy (SSRC): a single-institutionalprospectivestudy. SurgEndosc 27:2156–2162
- 16. Ramai D, Bhandari P, Facciorusso A, Barakat M, Pasisnichenko Y, Saghir S, Ambrosi A, Tartaglia N, Chandan S, Dhindsa B, Dhaliwal A, McDonough S, Adler DG. Real-World Experience of Intragastric Balloons for Obesity: Insights from the FDA Manufacturer and User Facility Device Experience (MAUDE) Database. ObesSurg. 2021 Jul;31(7):3360-3364. doi: 10.1007/s11695-021-05324-x. Epub 2021 Mar 9. PMID: 33687626.
- 17. Singhal R, Ludwig C, Rudge G, Gkoutos GV, Tahrani A, Mahawar K; GENEVA Collaborators, et al. 30-Day Morbidity and Mortality of Bariatric Surgery During the COVID-19 Pandemic: a Multinational Cohort Study of 7704 Patients from 42 Countries. Obes Surg. 2021 Oct;31(10):4272-4288. doi: 10.1007/s11695-021-05493-9. Epub 2021 Jul 30. PMID: 34328624; PMCID: PMC8323543.
- 18. Tartaglia N, Pavone G, Lizzi V, Vovola F, Tricarico F, Pacilli M, Ambrosi A. How emergency surgery has changed during the COVID-19 pandemic: A cohort study. Ann Med Surg (Lond). 2020 Dec 5;60:686-689. doi: 10.1016/j.amsu.2020.12.001. PMID: 33312562; PMCID: PMC7719013.
- 19. Rosenthal RJ, International Sleeve Gastrectomy Expert Panel, Diaz AA, et al. International sleeve gastrectomy expert panel consensus statement: best practice guidelines based on experience of >12,000 cases. SurgObesRelatDis. 2012;8(1):8–

- 20. Balagué C, Ruiz de Adana JC, Ibarzabal A, et al. Insights into the treatment of postsleeve gastrectomy leak: analysis of the results of 105 cases on a national register. SurgObesRelatDis. 2021;17(1):36–43.
- 21. Benedix F, Benedix DD, Knoll C, et al. Are there risk factors that increase the rate of staple line leakage in patients undergoing primary sleeve gastrectomy for morbid obesity? ObesSurg. 2014;24(10):1610–6.
- 22. Delle Monache S, Calgani A, Sanità P, et al. Adipose-derived stem cells sustain prolonged angiogenesis through leptin secretion. GrowthFactors. 2016;34(3–4):87–96. https://doi.org/10.1080/08977194.2016.1191481.
- 23. Parikh M, Issa R, McCrillis A, et al. Surgical strategies that may decrease leak after laparoscopic sleeve gastrectomy: a systematic review and metaanalysis of 9991 cases. AnnSurg. 2013;257(2): 231–7.
- 24. Aggarwal S, Bhattacharjee H, ChanderMisra M. Practice of routine intraoperative leak test during laparoscopic sleeve gastrectomy should not be discarded. SurgObesRelatDis. 2011;7(5):e24–5.
- 25. Degett TH, Andersen HS, Gögenur I. Indocyanine green fluorescence angiography for intraoperative assessment of gastrointestinal anastomotic perfusion: a systematic review of clinical trials. Langenbeck's Arch Surg. 2016;401(6):767–75. https://doi.org/10.1007/s00423-016-1400-9.
- 26. Di Furia M, Romano L, Salvatorelli A, Brandolin D, Lomanto D, Cianca G, Schietroma M, Carlei F, Giuliani A. Indocyanine Green FluorescentAngiographyDuringLaparoscopic Sleeve Gastrectomy: Preliminary Results. ObesSurg. 2019 Dec;29(12):3786-3790. doi: 10.1007/s11695-019-04085-y. PMID: 31290111.
- 27. Ortega CB, Guerron AD, Yoo JS. The Use of Fluorescence Angiography During Laparoscopic Sleeve Gastrectomy. JSLS. 2018 Apr-Jun;22(2):e2018.00005. doi: 10.4293/JSLS.2018.00005. PMID: 29950800; PMCID: PMC6016860.
- 28. Frattini F, Lavazza M, Mangano A, Amico F, Rausei S, Rovera F, Boni L, Dionigi G. Indocyanine green-enhancedfluorescence in laparoscopic sleeve gastrectomy.

- ObesSurg. 2015 May;25(5):949-50. doi: 10.1007/s11695-015-1640-8. PMID: 25736231.
- 29. Cianci P, Tartaglia N, Altamura A, Di Lascia A, Fersini A, Neri V, Ambrosi A. Cervical Esophagotomy for Foreign Body Extraction: A Case Report and Extensive Literature Review of the Last 20 Years. Am J Case Rep. 2018 Apr 5;19:400-405. doi: 10.12659/ajcr.908373. PMID: 29618719; PMCID: PMC5900799.
- 30. Cobianchi L, Dal Mas F, Massaro M, Fugazzola P, Coccolini F, Kluger Y, Leppäniemi A, Moore EE, Sartelli M, Angelos P, Catena F, Ansaloni L; Team Dynamics Study Group. Team dynamics in emergency surgery teams: results from a first international survey. World J Emerg Surg. 2021 Sep 16;16(1):47. doi: 10.1186/s13017-021-00389-6. Erratum in: World J Emerg Surg. 2021 Nov 1;16(1):55. PMID: 34530891; PMCID: PMC8443910.

Ethics approval and consent to participate: The ethics committee (DDG n. 363 del

25/10/2016 e s.m.i. DDG n. 318 del 14/06/2019) of our institution (PoliclinicoRiuniti)

approved the study.

All research methods were carried out in accordance with relevant guidelines and

regulations.

Written informed consent was obtained.

**Consent for publication:** Not Applicable.

**Availability of data and materials:** All data generated or analysed during this study are

included in this published article.

**Competing interests:** The authors declare no competing interests.

**Funding:** No funding

Authors' contributions:

GIOVANNA PAVONE and NICOLA TARTAGLIA performed the study conception

and design.

MARIO PACILLI, FRANCESCA MADDALENA and FABIO PETRUZZELLI

analysed and interpreted the data.

GENNARO MARTINES and MICHELE DE FAZIO contributed to acquisition of

the data.

ANTONIO AMBROSI revised the manuscript.

Figure 1a: Evaluation of perfusion of staple line of the stomach by using Indocyanine green test

Figure 1b: Intraoperative picture of the staple line of the stomach

Figure 2: Gastrografin swallow test

- Figure 3: The collection and the air pocket adjacent to the staple line at the upper stomach on the abdominal CT
- Figure 4: The endoscopic evidence of the gastric fistula
- Figure 5: Self-expanding covered prosthesis placed to exclude the fistula
- Figure 6: Control abdomen CT that shows a clear reduction of the intra-abdominal collection